CLINICAL TRIAL: NCT03217760
Title: Patient's Induced Stress and Young Practitioner's Induced Stress During Endodontic Therapy.
Brief Title: Stress Factors Induced by Patient and Young Clinicien During Endodontic Treatment
Acronym: STRESSENDO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: STRESSENDO (16.118)
Record Dates: First submitted 2017-06-20; First posted 2017-07-14 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Endodontic Treatment
Keywords: Induced stress, dental anxiety, endodontic treatment, salivary cortisol, cardiovascular parameters, pain, discomfort.
MeSH Terms: conditions — Pain | interventions — Endodontics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Salivary samples are collected during endodontic treatment to measure cortisol production during endodontic treatment. Cortisol is a hormone secreted from the adrenal cortex and dispersed to all body fluids (urine, serum, or saliva). A correlation between salivary cortisol levels and stress in dental procedure is noticed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: The main aim of the study is to examine the patient's induced stress during endodontic treatment in order to offer customised solutions to lessen stress. The other aims is also to evaluate the patient's pain and discomfort during endodontic treatment.
  Interventions: Other: VAS of stress; Other: CORAH scale; Other: HAD Scale; Other: Cardiovascular Parameters; Other: Cortisol Measurements; Other: Discomfort and Pain Experienced During Treatment; Other: Patient's preferences.
- Young dentists practitioners.: The other aims are to evaluate the young dentist's induced stress and to examine and compare the patient's induced stress and the young dentist's induced stress.
  Interventions: Procedure: Endodontic treatment; Other: VAS of stress; Other: HAD Scale; Other: Cardiovascular Parameters; Other: Cortisol Measurements; Other: student preferences.

INTERVENTIONS:
Procedure: Endodontic treatment — Endodontic treatment or root canal therapy is a sequence of treatment for the infected pulp of a tooth which results in the elimination of infection and the protection of the decontaminated tooth from future microbial invasion.
  Groups: Young dentists practitioners.
Other: VAS of stress — The VAS is a 10-cm scale without graduation on which subjects are asked to score the specific level of stress experienced from 0 (not stressed at all) to 10 (worst stress imaginable)
Other: CORAH scale — At the beginning of the treatment (T1), the patient is asked to complete a French version of the Corah Dental Anxiety scale (DAS).
  Groups: Patients
Other: HAD Scale — At the beginning of the treatment (T1), patients and students are asked to complete the Hospital Anxiety and Depression Scale (HAD Scale) which is presented as a reliable instrument for assessing clinically significant anxiety and depression.
Other: Cardiovascular Parameters — For each subject, the physiological indicators of stress (ie, heart rate [HR], systolic blood pressure [SBP], and diastolic blood pressure [DBP]) are monitored during each of the 6 steps.
Other: Cortisol Measurements — Salivary samples are collected during each of the 6 steps of endodontic treatment which are then stored at -20° before being sent to the laboratory to test cortisol levels .
Other: Discomfort and Pain Experienced During Treatment — Patients were asked to report the levels of discomfort and pain experienced during the 6 steps using the VAS and at the next visit for the final restoration.
  Groups: Patients
Other: Patient's preferences. — After the completion of each treatment patients will have to report whether they thought that they would have experienced as much pain, stress, or discomfort if they had received premedication before treatment.
  Groups: Patients
Other: student preferences. — When the treatment is complete the students are asked to report:
  1. his/her level of satisfaction with the course of treatment,
  2. whether he/she felt awkward faced with the patient's manifestations of stress, discomfort, or pain during the session
  3. whether he/she would have preferred that the patient had received sedative medication before the endodontic treatment.
  Groups: Young dentists practitioners.

SUMMARY:
The aim of this pilot study is to examine the patient's induced stress and the young dentist's induced stress, during endodontic treatment. This study is carried out using physiologic (cortisol measurement, arterial pressure and heart rate) and psychological data (VAS visual analog scale of stress, pain and discomfort, CORAH and HAD Scales) collected from patients of Brest University Dental Hospital at various stages of root canal treatment. The endodontic treatment is carried out under the usual standards and practices.

DETAILED DESCRIPTION:
Thirty patients and students are involved. All adult patients referred to the dental department for initial endodontic treatment are given the option of taking part, excluding those presenting cardiovascular disease or mental, psychiatric, or neuronal disease. Patients taking antihypertensive treatment, anxiolytics, sedatives, or neuroleptic drugs are also excluded from the study. Thirty dental students will conduct endodontic treatments according to the regular local procedures. No patient receives any sedative premedication.

The indicators of stress are monitored at 6 steps of endodontic treatment:

T1: preoperative rest; T2: local anaesthesia (4% articaïne hydrochloride with 1:200 000 epinephrine). T3: rubber-dam set-up T4: root canal instrumentation T5: root canal filling T6: postoperative rest

The main study criteria is the variation of stress:

At the 6 steps of the treatment and at the next visit for the final restoration, both subjects (patient and student) are asked to use a visual analog scale (VAS) to score the level of stress specifically induced by the endodontic treatment. The VAS is a 10-cm scale without graduation on which subjects are asked to score the specific level of stress experienced from 0 (not stressed at all) to 10 (worst stress imaginable). The VAS of stress has proven to be a valid tool that is highly sensitive to change.

Other study criteria:

- CORAH and HAD Scales At the beginning of the treatment (T1), the patient is asked to complete a French version of the Corah Dental Anxiety scale (DAS). This questionnaire consists of 4 parts: the results lead to the assessment of dental anxiety.

At the beginning of the treatment (T1), patients and students are asked to complete the Hospital Anxiety and Depression Scale (HAD Scale) which is presented as a reliable instrument for assessing clinically significant anxiety and depression in patients.

* Cardiovascular Parameters For each subject, the physiological indicators of stress (ie, heart rate [HR], systolic blood pressure [SBP], and diastolic blood pressure [DBP]) are monitored during each of the 6 steps.
* Cortisol Measurements A correlation between salivary cortisol level and stress in dental procedure was noticed .

Salivary samples are collected during each of the 6 steps of endodontic treatment which are then stored at -20° before being sent to the laboratory to test cortisol levels .

* Discomfort and Pain Experienced During Treatment Dental anxiety was found to have a direct relationship with pain perception (). Patients were asked to report the levels of discomfort and pain experienced during the 6 steps using the VAS and at the next visit for the final restoration.
* Patient and student preferences After the completion of each scale patients will have to report whether they thought that they would have experienced as much pain, stress, or discomfort if they had received premedication before treatment.

When the treatment is complete the students are asked to report:

1. his/her level of satisfaction with the course of treatment,
2. whether he/she felt awkward faced with the patient's manifestations of stress, discomfort, or pain during the session
3. whether he/she would have preferred that the patient had received sedative medication before the endodontic treatment.

The main aim of the study is to examine the patient's induced stress during endodontic treatment in order to offer customised solutions to lessen stress. The other aims are to evaluate the young dentist's induced stress, to examine and compare the patient's induced stress and the young dentist's induced stress, and to evaluate the patient's pain and discomfort during endodontic treatment.

The results of this observational study are to be used as a reference for future interventional studies to reduce stress during endodontic treatment. Techniques such as relaxation, hypnosis, acupuncture, distraction, music therapy, positive reinforcement, stop-signalling, and exposure-based treatments, "tell-show-do" are some solutions which could be initiated at the dentistry department of CHRU Brest.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years old
* Patients who need endodontic treatment
* Patients insured under the French social security system

Exclusion Criteria:

* Pregnant women
* Participants refusing to take part
* Patients not fluent in French.
* Patients who have certain diseases which do not allow interpretion of the cardiovascular outcomes (cardiac rhythm disorder, hypertension)
* Treatments or diseases which may have profound implications on stress modulation
* Certain diseases which affect cortisol levels: Cushing, Addison, obesity (body mass index (BMI) > 30 kg/m²), schizophrenia, personality and behaviour disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients and students were needed.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
The main study criteria is the variation of stress. | At the 6 steps of the treatment and at the next visit for the final restoration : up to 15 days
  At the 6 steps of the treatment and at the next visit for the final restoration, both subjects (patient and student) are asked to use a visual analog scale (VAS) to score the level of stress specifically induced by the endodontic treatment. The VAS is a 10-cm scale without graduation on which subjects are asked to score the specific level of stress experienced from 0 (not stressed at all) to 10 (worst stress imaginable). The VAS of stress has proven to be a valid tool that is highly sensitive to change.

SECONDARY OUTCOMES:
CORAH . | At the beginning of the treatment (T1) : one day
  At the beginning of the treatment (T1), the patient is asked to complete a French version of the Corah Dental Anxiety scale (DAS). This questionnaire consists of 4 parts: the results lead to the assessment of dental anxiety.
  At the beginning of the treatment (T1), patients and students are asked to complete the Hospital Anxiety and Depression Scale (HAD Scale) which is presented as a reliable instrument for assessing clinically significant anxiety and depression in patients.
HAD Scales. | At the beginning of the treatment (T1) : one day
  At the beginning of the treatment (T1), the patient is asked to complete a French version of the Corah Dental Anxiety scale (DAS). This questionnaire consists of 4 parts: the results lead to the assessment of dental anxiety.
  At the beginning of the treatment (T1), patients and students are asked to complete the Hospital Anxiety and Depression Scale (HAD Scale) which is presented as a reliable instrument for assessing clinically significant anxiety and depression in patients.
Cardiovascular Parameters | During endodontie treatment (one day) and at the next visit for the final restoration (15 days after).
  For each subject, the physiological indicators of stress (heart rate [HR]) are monitored during each of the 6 steps.
Cardiovascular Parameters | During endodontie treatment (one day) and at the next visit for the final restoration (15 days after)
  For each subject, the physiological indicators of stress (systolic blood pressure [SBP]) are monitored during each of the 6 steps.
Cardiovascular Parameters | During endodontie treatment (one day) and at the next visit for the final restoration (15 days after)
  For each subject, the physiological indicators of stress (diastolic blood pressure [DBP]) are monitored during each of the 6 steps.
Cortisol Measurements | During endodontic treatment (one day).
  A correlation between salivary cortisol level and stress in dental procedure was noticed.
  Salivary samples are collected during each of the 6 steps of endodontic treatment which are then stored at -20° before being sent to the laboratory to test cortisol levels .
Discomfort and Pain Experienced During Treatment | During endodontic treatment (one day) and at the next visit for the final restoration (15 days after).
  Dental anxiety was found to have a direct relationship with pain perception ((Sathorn et al., 2008)). Patients were asked to report the levels of discomfort and pain experienced during the 6 steps using the VAS and at the next visit for the final restoration.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France